CLINICAL TRIAL: NCT01678443
Title: A Phase I Study Evaluating Escalating Doses of 90Y-BC8-DOTA (Anti-CD45) Antibody Followed by Autologous Stem Cell Transplantation for Relapsed or Refractory Lymphoid Malignancies
Brief Title: Monoclonal Antibody Therapy Before Stem Cell Transplant in Treating Patients With Relapsed or Refractory Lymphoid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to low accrual.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Gopal, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2361.00; NCI-2012-01505 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2361.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P01CA044991 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Indium; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (yttrium-90 anti-CD45 monoclonal antibody BC8) (Experimental): Patients receive indium-111 anti-CD45 monoclonal antibody BC8 IV on day -28 and (if necessary) day -21. Patients receive yttrium-90 anti-CD45 monoclonal antibody BC8 IV on day -28, -14, and -13. Patients then undergo autologous peripheral blood stem cell transplantation on day 0.
  Interventions: Biological: indium In 111 anti-CD45 monoclonal antibody BC8; Radiation: yttrium Y 90 anti-CD45 monoclonal antibody BC8; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: indium In 111 anti-CD45 monoclonal antibody BC8 — Given IV
  Other Names: In 111 MOAB BC8; In 111 monoclonal antibody BC8; In111 MOAB BC8; indium In 111 MOAB BC8
Radiation: yttrium Y 90 anti-CD45 monoclonal antibody BC8 — Given IV
  Other Names: 90Y anti-CD45 MAb BC8; 90Y anti-CD45 MoAb BC8
Procedure: peripheral blood stem cell transplantation — Undergo autologous peripheral blood stem cell transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell

SUMMARY:
This phase I trial studies the side effects and best dose of monoclonal antibody therapy before stem cell transplant in treating patients with relapsed or refractory lymphoid malignancies. Radiolabeled monoclonal antibodies, such as yttrium-90 anti-CD45 monoclonal antibody BC8, can find cancer cells and carry cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving radiolabeled monoclonal antibody before a stem cell transplant may be an effective treatment for relapsed or refractory lymphoid malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximally tolerated dose (MTD) of 90Y-BC8-DOTA (anti-cluster of differentiation [CD]45) (yttrium-90 anti-CD45 monoclonal antibody BC8) that can be delivered prior to autologous stem cell transplantation for patients with relapsed/refractory B-cell non-Hodgkin lymphoma (B-NHL), T-cell NHL (T-NHL), and Hodgkin lymphoma (HL).

SECONDARY OBJECTIVES:

I. To optimize the protein dose (antibody [Ab]) to deliver a favorable biodistribution in the majority of patients.

II. To describe the impact of rituximab concentrations, B-cell depletion, and disease burden on CD20 and CD45 targeting.

III. To describe response rates and remission durations in relapsed B-NHL, T-NHL, and HL following administration of myeloablative doses of 90Y-BC8-DOTA prior to autologous stem cell transplant (ASCT).

IV. To assess the correlation of lymphoma biomarkers with outcomes.

OUTLINE: This is a dose-escalation study of yttrium-90 anti-CD45 monoclonal antibody BC8.

Patients receive indium-111 anti-CD45 monoclonal antibody BC8 intravenously (IV) on day -28 and (if necessary) day -21 to evaluate the antibody's biodistribution. Patients then receive yttrium-90 anti-CD45 monoclonal antibody BC8 IV on day -14. Patients then undergo autologous peripheral blood stem cell transplantation on day 0.

After completion of study treatment, patients are followed up at 3, 6, and 12 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of B-NHL, T-NHL, or HL; only patients with classical HL must have documented histologic demonstration of CD45+ cells adjacent to the Reed Sternberg cells; patients must have received at least one prior standard systemic therapy with documented recurrent or refractory disease; patients with mantle cell lymphoma (MCL), T-NHL, or other high-risk malignancies may be enrolled/transplanted in complete remission (CR)/first partial remission (PR1)
* Creatinine < 2.0
* Bilirubin < 1.5 mg/dL
* All patients eligible for therapeutic study must have a minimum of >= 2 x 10^6 CD34/kg autologous hematopoietic stem cells harvested and cryopreserved
* Patients must have an expected survival of > 60 days and must be free of major infection
* Patients are preferred to have either a tumor mass amenable to core needle biopsy during the dosimetry phase, or a measurable tumor mass with at least one site of involvement measuring 2.5 cm in largest dimension on computed tomography (CT) imaging for purposes of planar and/or single-photon emission computed tomography (SPECT)/CT tumor dosimetry

Exclusion Criteria:

* Circulating human anti-mouse antibody (HAMA), to be determined before each infusion
* Systemic anti-lymphoma therapy given in the previous 30 days before the scheduled therapy dose with the exception of rituximab
* Inability to understand or give an informed consent
* Lymphoma involving the central nervous system
* Other serious medical conditions considered to represent contraindications to ASCT (e.g., abnormally decreased cardiac ejection fraction, diffusion capacity of the lung for carbon monoxide [DLCO] < 50% predicted, acquired immune deficiency syndrome [AIDS], etc.)
* Known human immunodeficiency virus (HIV) seropositivity
* Pregnancy or breast feeding
* Prior allogeneic bone marrow or stem cell transplant
* Prior autologous bone marrow or stem cell transplant within 1 year of enrollment
* Prior radiation therapy (RT) > 20 Gray (Gy) to a critical organ within 1 year of enrollment
* Southwest Oncology Group (SWOG) performance status >= 2.0
* Patients with relapsed diffuse large B-cell lymphoma (DLBCL) or HL that have achieved a positron emission tomography (PET)-negative CR following first salvage chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 1999-09-01 (Actual); Primary Completion 2013-09-21 (Actual); Study Completion 2018-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Yttrium-90 Anti-CD45 Monoclonal Antibody BC8)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Yttrium-90 Anti-CD45 Monoclonal Antibody BC8)
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities (DLT) of Yttrium-90 Anti-CD45
Description: A DLT (dose limiting toxicity) is defined as a therapy-related grade III or IV Bearman (transplant) toxicity within 30 days of transplant.
Time Frame: Up to 30 days after receiving study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Yttrium-90 Anti-CD45 Monoclonal Antibody BC8)
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Overall Response Rate
Time Frame: Up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Yttrium-90 Anti-CD45 Monoclonal Antibody BC8)
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Overall Survival
Time Frame: Up to 6 years
Measure: Mean (Full Range); unit: days
Arm/Group | Treatment (Yttrium-90 Anti-CD45 Monoclonal Antibody BC8)
Number analyzed (Participants) | 2
days | 750.5 [243 to 1258]

4. Secondary Outcome: Progression-free Survival
Time Frame: Up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Yttrium-90 Anti-CD45 Monoclonal Antibody BC8)
Number analyzed (Participants) | 2
Participants | 0

5. Secondary Outcome: Tumor to Normal Organ Ratios
Description: Derived from dosimetry estimates coupled with the absorbed dose to normal organs based on the administered activity of 90Y.
Time Frame: Up to 6 years
Population: This outcome measure was not done. Only two patients were enrolled before the study was closed early. Tumor to normal organ ratios was not determined due to small sample size.
Arm/Group | Treatment (Yttrium-90 Anti-CD45 Monoclonal Antibody BC8)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs will be monitored and recorded in study-specific case report forms (CRFs) from the time of first exposure to the investigational product in this study (i.e., the start of the first dosimetry infusion) through day +30 post transplant or through discharge prior to that date from the SCCA system to care of the patient's primary physician
Arm/Group | Treatment (Yttrium-90 Anti-CD45 Monoclonal Antibody BC8)
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Yttrium-90 Anti-CD45 Monoclonal Antibody BC8) (N=2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was closed when replaced by a new study adding chemotherapy to this regimen

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes